CLINICAL TRIAL: NCT00792896
Title: A Longitudinal Study That Assessed the Effectiveness of Intervention Toward
Brief Title: Intervention Toward Truth-Telling and Advanced Directives in the Patient With Advanced or Metastatic Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Responsible Party: 1, Jen-Ai Road Section 1, Taipei, Taiwan, Department of Nursing
Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 200803051R
Record Dates: First submitted 2008-11-16; First posted 2008-11-18 (Estimated); Last update posted 2008-11-18 (Estimated); Status verified 2008-05

CONDITIONS: Advanced Cancer; Metastatic Cancer
MeSH Terms: conditions — Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Family conference + education materials
  Interventions: Behavioral: family conference
- 2 (No Intervention): education materials

INTERVENTIONS:
Behavioral: family conference — family conference
  Arms: 1

SUMMARY:
Family usually had a lot of burden to tell the truth to patients. The purpose of this study is to assess the effect of education materials and family conference for advanced cancer patients and family.

ELIGIBILITY:
Inclusion Criteria:

* advanced or metastatic cancer patients
* more than 20 years old
* clear consciousness and be able to communicate

Exclusion Criteria:

* refuse to know the statement of himself/herself disease

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2008-05; Primary Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
Questionnaires | before and 1 week after the intervention

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan